CLINICAL TRIAL: NCT00006411
Title: Cornea Donor Study: The Effect of Donor Age on Penetrating Keratoplasty for Endothelial Disease
Brief Title: Cornea Donor Study
Acronym: CDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: Eye Bank Association of America (Other); Bausch & Lomb Incorporated (Industry); Tissue Banks International (Unknown); Vision Share, Inc. (Industry); San Diego Eye Bank (Other); The Cornea Society (Other); Katena Products, Inc. (Industry); ViroMed Laboratories, Inc. (Industry); Midwest Eye Banks (Other); Konan Medical, Inc. (Industry); Eye Bank for Sight Restoration (Unknown); SightLife (Other); Sight Society of Northeastern New York (Lions Eye Bank of Albany) (Unknown); Lions Eye Bank of Oregon (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NEI-80; 5U10EY012358 (NIH); 3U10EY012358-11S1 (NIH); 5U10EY012728 (NIH)
Record Dates: First submitted 2000-10-13; First posted 2000-10-16 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2018-08

CONDITIONS: Corneal Disease; Fuch's Dystrophy; Pseudophakic Corneal Edema
Keywords: cornea transplant; corneal endothelial cell density; moderate risk corneal diseases; corneal transplantation
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): cornea assigned from donor age group <66.0 years
  Interventions: Other: corneas assigned by donor age group
- 2 (Active Comparator): cornea assigned from donor age group >= 66.0 years
  Interventions: Other: corneas assigned by donor age group

INTERVENTIONS:
Other: corneas assigned by donor age group — A web-based computer program was used to select and assign a cornea by donor age group from those available at the eye bank that met the study eligibility criteria. The program randomly selected a cornea based on a two-level minimization procedure which attempted first to balance for each surgeon the number of corneas from donors >=66 and <66 years old and then, when possible, to balance among age subgroups of 10-35, 36-50, 51-65, 66-70, and 71-75 years. The assignment was made without regard to recipient age or any other subject characteristics.

SUMMARY:
The Cornea Donor Study (CDS) was designed as a prospective cohort study with the following objectives:

To determine whether the graft-failure rate over a 5-year follow-up period following corneal transplantation is the same when using corneal tissue from donors older than 65 years of age compared with tissue from younger donors.

To assess the relationship between donor/recipient ABO blood type compatibility and graft failure due to rejection.

To assess corneal endothelial cell density as an indicator of the health of the cornea and as a alternate outcome measure (in an optional Specular Microscopy Ancillary Study).

DETAILED DESCRIPTION:
The study enrolled 1101 subjects with a corneal disease considered to be at moderate risk for failure (principally Fuchs' dystrophy and pseudophakic corneal edema). A donor cornea meeting the following criteria was assigned to the subject by one of 43 participating eye banks:

* donor age 10 to 75 years
* endothelial cell count 2300 to 3300
* tissue quality very good to excellent
* death to preservation time <12 hrs if body refrigerated or eyes on ice and <8 hrs if not
* death to surgery time <5 days

The cornea surgeon (investigator) and patient were masked to donor age and characteristics of the donor cornea. Preoperative management, surgical technique, and postoperative care, including prescription of medications, were provided according to each investigator's customary routine. The follow-up visit schedule for the initial six months was left to each investigator's discretion and after this time the minimum follow-up visit schedule included a visit between six and 12 months and then one visit every 12 months through five years. The primary study outcome was graft survival at five years. The definition of graft failure, based on the definition used in Collaborative Corneal Transplantation Studies, was a regraft or, in the absence of regraft, a cloudy cornea in which there was loss of central graft clarity sufficient to compromise vision for a minimum of three consecutive months. Follow-up in the initial phase of the study continued for five years unless the patient had a regraft of the study eye.

For the ABO compatibility study, the ABO blood type of both the donor and recipient were determined in order to compare the rate of graft failure for ABO-compatible cases with the rate for ABO-incompatible cases.

For the Specular Microscopy Ancillary Study, endothelial cell counts were determined from specular images by a central reading center, and the relationship of the cell counts to donor age were assessed. In the initial phase of the study, specular images were obtained at 6 months, and then annually through five years post-transplant.

Five-year follow up was completed in November 2007. The 5-year cumulative probability of success was 86%: 86% in the <66.0 year donor age group and 86% in the >=66.0 year donor age group (difference = 0%, upper limit of one-sided 95% confidence interval = 4%). Adjusting for baseline endothelial cell density had no appreciable effect on these results. In a statistical model with donor age as a continuous variable, there was not a significant relationship between donor age and outcome (P=0.11). Three graft failures were due to primary donor failure, 8 to uncorrectable refractive error, 48 to graft rejection, 46 to endothelial decompensation, and 30 to other causes. At least one probable or definite graft rejection episode preceded graft failure in 23 of the 46 failures attributed to endothelial decompensation (4 definite and 19 probable) and in 18 of the 30 failures attributed to other causes (4 definite and 14 probable). The distribution of causes of failure between the donor age groups did not substantially differ.

Although the 5-year results indicated no difference in the success rate of moderate-risk transplants according to donor age, results from the SMAS indicated that among the successful cases, there was a slight association between donor age and endothelial cell loss, with the cell loss after 5 years being slightly lower in corneas from younger donors (r adjusted for baseline endothelial cell density = -0.19, 95% confidence interval -0.29 to -0.08). Whether this slight association between cell loss and donor age is of clinical importance is not known. Of perhaps even greater importance, however, was the finding that irrespective of donor age, endothelial cell loss was substantial over the first five years after transplant even when the graft had been successful. Half of the successful cases experienced a cell loss of 70% or more, and at five years more than half had an endothelial cell density <800 cells/mm2.

Patients in the CDS continued in annual follow up through 2012 in order to to determine the overall 10-year survival rate for moderate risk grafts and to determine whether the graft-failure rate is related to donor age. Additional objectives included determining the value of endothelial cell density in predicting graft failure and evaluating donor and recipient characteristics that may be predictive of late graft failure. All CDS subjects who were active at the 5-year exam were eligible for the extended follow-up phase.

As part of the Specular Microscopy Ancillary Study, follow-up images were obtained during the extended follow-up phase at 7-8 years and again at 10-years. The same procedures used during the first 5 years were followed for the grading of the 7-8 year and 10-year images.

ELIGIBILITY:
Inclusion

1. Age range 40-80 years
2. Corneal disease: Presence of a condition associated with endothelial dysfunction, including pseudophakic/aphakic corneal edema, Fuchs' dystrophy, posterior polymorphous dystrophy, interstitial keratitis (nonherpetic) or perforating corneal injury
3. Willingness to be followed for 5 years and life expectancy at least 5 years (in investigator's judgement)

Exclusion

1. Patients are to be excluded when there is:

   * a high risk of graft failure, including failed prior penetrating keratoplasty in the eye to be transplanted, chemical burns or other significant cicatricial conjunctivitis (ocular surface disease), herpes simplex/zoster, temporary keratoprosthesis, iridocorneal endothelial syndrome or any corneal condition in which there are two or more quadrants of stromal neovascularization

     * A quadrant is considered vascularized if there is at least one patent stromal vessel >2.0 mm in length crossing the limbus within a quadrant. Two quadrants are considered vascularized if there are at least two stromal vessels 90º or more apart. Enrollment will be restricted to no more than 20% of the total cohort having stromal neovascularization.
     * Patients should be excluded if there are PAS or other abnormalities that, in the view of the investigator, place the patient at high risk for graft failure.
   * a very high probability of success including keratoconus, stromal dystrophies, stromal scars without edema or post-refractive surgery with healthy endothelium
2. Uncontrolled glaucoma or prior filtering surgery with placement of a shunt in the eye to be grafted (Note: eyes requiring a filtering procedure combined with the PK are considered to have uncontrolled glaucoma and are ineligible. Eyes which have undergone filtering surgery (without a shunt) in which glaucoma is currently considered under control are eligible)
3. Uncontrolled uveitis in the eye to be grafted
4. Fellow eye visual acuity <20/200
5. Fellow eye already included in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1090 (Actual)
Dates: Start 2000-01-10 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Holland, MD, Study Chair — University of Cincinnati and Cincinnati Eye Institute; Mark J Mannis, MD, Study Chair — University of California, Davis; Roy W Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research; Jonathan H Lass, MD, Principal Investigator — (PI of Specular Microscopy Ancillary Study), Case Western Reserve University and University Hospitals Case Medical Center
Locations (1):
- Jaeb Center for Health Research, Inc., Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Public dataset access: http://cds.jaeb.org/Studies.aspx?RecID=185

REFERENCES:
- [Background] Beck RW, Gal RL, Mannis MJ, Holland EJ, Cavanagh HD, Foulks GN, Heck EL, Lindquist T, Macsai MS, Smith RE, Stark WJ, Stulting RD, Sugar J. Is donor age an important determinant of graft survival? Cornea. 1999 Sep;18(5):503-10. doi: 10.1097/00003226-199909000-00001. No abstract available. PMID 10487423
- [Background] Powe A, Gal RL, Beck RW, Mannis MJ, Holland EJ on behalf of the Cornea Donor Study Investigator Group. The Cornea Donor Study. Vision Pan-America 2009; 8:134-137.
- [Result] Sugar A, Gal RL, Beck rW, Ruedy KJ, Blanton CL, Feder RS, Hardten DR, Holland EJ, Lass JH, Mannis MJ, O'Keefe MB; Cornea Donor Study Group. Baseline donor characteristics in the Cornea Donor Study. Cornea. 2005 May;24(4):389-96. doi: 10.1097/01.ico.0000151503.26695.f0. PMID 15829793
- [Result] Lass JH, Gal RL, Ruedy KJ, Benetz BA, Beck RW, Baratz KH, Holland EJ, Kalajian A, Kollman C, Manning FJ, Mannis MJ, McCoy K, Montoya M, Stulting D, Xing D; Cornea Donor Study Group. An evaluation of image quality and accuracy of eye bank measurement of donor cornea endothelial cell density in the Specular Microscopy Ancillary Study. Ophthalmology. 2005 Mar;112(3):431-40. doi: 10.1016/j.ophtha.2004.10.045. PMID 15745770
- [Result] Mannis MJ, Holland EJ, Beck RW, Belin MW, Goldberg MA, Gal RL, Kalajian AD, Kenyon KR, Kollman C, Ruedy KJ, Smith P, Sugar J, Stark WJ; Cornea Donor Study Group. Clinical profile and early surgical complications in the Cornea Donor Study. Cornea. 2006 Feb;25(2):164-70. doi: 10.1097/01.ico.0000164832.69668.4b. PMID 16371775
- [Result] Benetz BA, Gal RL, Ruedy KJ, Rice C, Beck RW, Kalajian AD, Lass JH; Cornea Donor Study Group. Specular microscopy ancillary study methods for donor endothelial cell density determination of Cornea Donor Study images. Curr Eye Res. 2006 Apr;31(4):319-27. doi: 10.1080/02713680500536738. PMID 16603465
- [Result] Cornea Donor Study Investigator Group; gal RL, Dontchev M, Beck RW, Mannis MJ, Holland EJ, Kollman C, Dunn SP, Heck EL, Lass JH, Montoya MM, Schultze RL, Stulting RD, Sugar A, Sugar J, Tennant B, Verdier DD. The effect of donor age on corneal transplantation outcome results of the cornea donor study. Ophthalmology. 2008 Apr;115(4):620-626.e6. doi: 10.1016/j.ophtha.2008.01.003. PMID 18387407
- [Result] Cornea Donor Study Investigator Group; Lass JH, Gal RL, Dontchev M, Beck RW, Kollman C, Dunn SP, Heck E, Holland EJ, Mannis MJ, Montoya MM, Schultze RL, Stulting RD, Sugar A, Sugar J, Tennant B, Verdier DD. Donor age and corneal endothelial cell loss 5 years after successful corneal transplantation. Specular microscopy ancillary study results. Ophthalmology. 2008 Apr;115(4):627-632.e8. doi: 10.1016/j.ophtha.2008.01.004. PMID 18387408
- [Result] Sugar A, Tanner JP, Dontchev M, Tennant B, Schultze RL, Dunn SP, Lindquist TD, Gal RL, Beck RW, Kollman C, Mannis MJ, Holland EJ; Cornea Donor Study Investigator Group. Recipient risk factors for graft failure in the cornea donor study. Ophthalmology. 2009 Jun;116(6):1023-8. doi: 10.1016/j.ophtha.2008.12.050. Epub 2009 Apr 23. PMID 19395036
- [Result] Sugar J, Montoya M, Dontchev M, Tanner JP, Beck R, Gal R, Gallagher S, Gaster R, Heck E, Holland EJ, Kollman C, Malling J, Mannis MJ, Woody J; Group Cornea Donor Study Investigator Group. Donor risk factors for graft failure in the cornea donor study. Cornea. 2009 Oct;28(9):981-5. doi: 10.1097/ICO.0b013e3181a0a3e6. PMID 19724216
- [Result] Dunn SP, Stark WJ, Stulting RD, Lass JH, Sugar A, Pavilack MA, Smith PW, Tanner JP, Dontchev M, Gal RL, Beck RW, Kollman C, Mannis MJ, Holland EJ; Cornea Donor Study Investigator Group. The effect of ABO blood incompatibility on corneal transplant failure in conditions with low-risk of graft rejection. Am J Ophthalmol. 2009 Mar;147(3):432-438.e3. doi: 10.1016/j.ajo.2008.09.021. Epub 2008 Dec 4. PMID 19056078
- [Result] Lass JH, Sugar A, Benetz BA, Beck RW, Dontchev M, Gal RL, Kollman C, Gross R, Heck E, Holland EJ, Mannis MJ, Raber I, Stark W, Stulting RD; Cornea Donor Study Investigator Group. Endothelial cell density to predict endothelial graft failure after penetrating keratoplasty. Arch Ophthalmol. 2010 Jan;128(1):63-9. doi: 10.1001/archophthalmol.2010.128.63. PMID 20065219
- [Result] Lass JH, Beck RW, Benetz BA, Dontchev M, Gal RL, Holland EJ, Kollman C, Mannis MJ, Price F Jr, Raber I, Stark W, Stulting RD, Sugar A; Cornea Donor Study Investigator Group. Baseline factors related to endothelial cell loss following penetrating keratoplasty. Arch Ophthalmol. 2011 Sep;129(9):1149-54. doi: 10.1001/archophthalmol.2011.102. Epub 2011 May 9. PMID 21555600
- [Result] Stulting RD, Sugar A, Beck R, Belin M, Dontchev M, Feder RS, Gal RL, Holland EJ, Kollman C, Mannis MJ, Price F Jr, Stark W, Verdier DD; Cornea Donor Study Investigator Group. Effect of donor and recipient factors on corneal graft rejection. Cornea. 2012 Oct;31(10):1141-7. doi: 10.1097/ICO.0b013e31823f77f5. PMID 22488114
- [Result] Sugar A, Montoya MM, Beck R, Cowden JW, Dontchev M, Gal RL, Kollman C, Malling J, Mannis MJ, Tennant B; Cornea Donor Study Investigator Group. Impact of the cornea donor study on acceptance of corneas from older donors. Cornea. 2012 Dec;31(12):1441-5. doi: 10.1097/ICO.0b013e31823f7550. PMID 22262218
- [Result] Verdier DD, Sugar A, Baratz K, Beck R, Dontchev M, Dunn S, Gal RL, Holland EJ, Kollman C, Lass JH, Mannis MJ, Penta J; Cornea Donor Study Investigator Group. Corneal thickness as a predictor of corneal transplant outcome. Cornea. 2013 Jun;32(6):729-36. doi: 10.1097/ICO.0b013e31827b14c7. PMID 23343949
- [Result] Benetz BA, Lass JH, Gal RL, Sugar A, Menegay H, Dontchev M, Kollman C, Beck RW, Mannis MJ, Holland EJ, Gorovoy M, Hannush SB, Bokosky JE, Caudill JW; Cornea Donor Study Investigator Group. Endothelial morphometric measures to predict endothelial graft failure after penetrating keratoplasty. JAMA Ophthalmol. 2013 May;131(5):601-608. doi: 10.1001/jamaophthalmol.2013.1693. PMID 23493999
- [Result] Writing Committee for the Cornea Donor Study Research Group; Mannis MJ, Holland EJ, Gal RL, Dontchev M, Kollman C, Raghinaru D, Dunn SP, Schultze RL, Verdier DD, Lass JH, Raber IM, Sugar J, Gorovoy MS, Sugar A, Stulting RD, Montoya MM, Penta JG, Benetz BA, Beck RW. The effect of donor age on penetrating keratoplasty for endothelial disease: graft survival after 10 years in the Cornea Donor Study. Ophthalmology. 2013 Dec;120(12):2419-2427. doi: 10.1016/j.ophtha.2013.08.026. PMID 24246825
- [Result] Writing Committee for the Cornea Donor Study Research Group; Lass JH, Benetz BA, Gal RL, Kollman C, Raghinaru D, Dontchev M, Mannis MJ, Holland EJ, Chow C, McCoy K, Price FW Jr, Sugar A, Verdier DD, Beck RW. Donor age and factors related to endothelial cell loss 10 years after penetrating keratoplasty: Specular Microscopy Ancillary Study. Ophthalmology. 2013 Dec;120(12):2428-2435. doi: 10.1016/j.ophtha.2013.08.044. PMID 24246826
- [Result] Dunn SP, Gal RL, Kollman C, Raghinaru D, Dontchev M, Blanton CL, Holland EJ, Lass JH, Kenyon KR, Mannis MJ, Mian SI, Rapuano CJ, Stark WJ, Beck RW; Writing Committee for the Cornea Donor Study Research Group. Corneal graft rejection 10 years after penetrating keratoplasty in the cornea donor study. Cornea. 2014 Oct;33(10):1003-9. doi: 10.1097/ICO.0000000000000212. PMID 25119961
- [Result] Riddlesworth TD, Kollman C, Lass JH, Patel SV, Stulting RD, Benetz BA, Gal RL, Beck RW. A mathematical model to predict endothelial cell density following penetrating keratoplasty with selective dropout from graft failure. Invest Ophthalmol Vis Sci. 2014 Nov 25;55(12):8409-15. doi: 10.1167/iovs.14-15683. PMID 25425307
- [Result] Writing Committee for the Cornea Donor Study Research Group; Sugar A, Gal RL, Kollman C, Raghinaru D, Dontchev M, Croasdale CR, Feder RS, Holland EJ, Lass JH, Macy JI, Mannis MJ, Smith PW, Soukiasian SH, Beck RW. Factors associated with corneal graft survival in the cornea donor study. JAMA Ophthalmol. 2015 Mar;133(3):246-54. doi: 10.1001/jamaophthalmol.2014.3923. PMID 25322173
- [Result] Lass JH, Riddlesworth TD, Gal RL, Kollman C, Benetz BA, Price FW Jr, Sugar A, Terry MA, Soper M, Beck RW; Cornea Donor Study Research Group. The effect of donor diabetes history on graft failure and endothelial cell density 10 years after penetrating keratoplasty. Ophthalmology. 2015 Mar;122(3):448-56. doi: 10.1016/j.ophtha.2014.09.012. Epub 2014 Nov 15. PMID 25439611

RESULTS

PARTICIPANT FLOW:
Groups:
- Cornea Assigned From Donor Age Group <66.0 Years: cornea assigned from donor age group <66.0 years
  corneas assigned by donor age group: A web-based computer program was used to select and assign a cornea by donor age group from those available at the eye bank that met the study eligibility criteria. The program randomly selected a cornea based on a two-level minimization procedure which attempted first to balance for each surgeon the number of corneas from donors >=66 and <66 years old and then, when possible, to balance among age subgroups of 10-35, 36-50, 51-65, 66-70, and 71-75 years. The assignment was made without regard to recipient age or any other subject characteristics.
- Cornea Assigned From Donor Age Group >= 66.0 Years: cornea assigned from donor age group >= 66.0 years
  corneas assigned by donor age group: A web-based computer program was used to select and assign a cornea by donor age group from those available at the eye bank that met the study eligibility criteria. The program randomly selected a cornea based on a two-level minimization procedure which attempted first to balance for each surgeon the number of corneas from donors >=66 and <66 years old and then, when possible, to balance among age subgroups of 10-35, 36-50, 51-65, 66-70, and 71-75 years. The assignment was made without regard to recipient age or any other subject characteristics.
Period: Overall Study
Arm/Group | Cornea Assigned From Donor Age Group <66.0 Years | Cornea Assigned From Donor Age Group >= 66.0 Years
Started | 707 | 383
Completed | 707 | 383
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cornea Assigned From Donor Age Group <66.0 Years | Cornea Assigned From Donor Age Group >= 66.0 Years | Total
Number analyzed (Participants) | 707 | 383 | 1090
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9) | 71 (8) | 70 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 445 | 252 | 697
  Male | 262 | 131 | 393

OUTCOME MEASURES:

1. Primary Outcome: Graft Failure
Description: # eyes with graft failure, defined as a regraft or a cloudy cornea that was sufficiently opaque as to compromise vision for a minimum of three consecutive months. Only one eye per participant was included in the study.
Time Frame: Baseline to 10 Years of Follow Up
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | Cornea Assigned From Donor Age Group <66.0 Years | Cornea Assigned From Donor Age Group >= 66.0 Years
Number analyzed (Participants) | 707 | 383
Number analyzed (eyes) | 707 | 383
participants | 142 | 82

2. Secondary Outcome: Endothelial Cell Density (ECD)
Description: ECD (cells/mm2)was measured on a subset of the overall Cornea Donor Study cohort who participated in the Specular Microscopy Ancillary Study
Time Frame: 10 year ECD
Population: Of 1,090 eligible participants enrolled in the CDS, the SMAS included 609. A gradable endothelial image at 10 years was available for 176 participants. Among the other 433 participants, 105 had a graft failure, 100 died, 103 completed less than 10 years of CDS follow up, and 125 did not have a 10-year image for other reasons.
Measure: Median (Inter-Quartile Range); unit: ECD (cells/mm2)
Arm/Group | Cornea Assigned From Donor Age Group <66.0 Years | Cornea Assigned From Donor Age Group >= 66.0 Years
Number analyzed (Participants) | 125 | 51
ECD (cells/mm2) | 628 [522 to 850] | 550 [483 to 694]

ADVERSE EVENTS:
Arm/Group | Cornea Assigned From Donor Age Group <66.0 Years | Cornea Assigned From Donor Age Group >= 66.0 Years
Serious Adverse Events (participants affected / at risk) | 0/707 | 0/383
Other Adverse Events (participants affected / at risk) | 0/707 | 0/383

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No